CLINICAL TRIAL: NCT01232790
Title: A Pilot Trial of Acute N-Acetylcysteine Effects on Working Memory and Other Cognitive Functions in Schizophrenia
Acronym: NAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0904005039; M131976 (Other Grant/Funding Number: NARSAD)
Record Dates: First submitted 2010-02-25; First posted 2010-11-02 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; working memory; N-Acetylcysteine
MeSH Terms: conditions — Schizophrenia | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Intervention/Placebo (Experimental): Group A first receives the commercially available sustained release form of N-acetylcysteine, then the matching placebo capsules both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days).
  Interventions: Dietary Supplement: N-Acetylcysteine
- Group B: Placebo/Intervention (Placebo Comparator): Group B first receives the placebo and then receives a commercially available sustained release form of N-Acetylcysteine. In each arm, the capsules are both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: N-Acetylcysteine — N-acetylcysteine 1200mg bid for 3 days
  Arms: Group A: Intervention/Placebo
Drug: Placebo — Placebo
  Arms: Group B: Placebo/Intervention

SUMMARY:
The purpose of this study is to evaluate the effects of the amino acid supplement N-Acetylcysteine versus placebo on working memory and other cognitive functions in persons with a diagnosis of schizophrenia.

DETAILED DESCRIPTION:
Working memory impairment in Schizophrenia is produced by deficiencies of feedback inhibition of glutamate release, due to low cysteine-glutamate antiporter activity. Because of this mechanism, we are interested in whether acute administration of N-Acetylcysteine will improve performance of patients with schizophrenia on a battery of cognitive tasks utilized to test working memory and other cognitive domains, versus placebo. This pilot study will utilize a randomized, double blind, placebo controlled, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between 18-60
* Meet Diagnostic and Statistical Manual-IV (DSM) criteria for schizophrenia
* Be on a stable dose of antipsychotic medication for at least 1 month
* Be deemed clinically stable for 3 months by the regular clinical staff

Exclusion Criteria:

* Current substance or alcohol abuse
* Pregnancy
* Clozapine treatment
* Known sensitivity to sulphur containing compounds
* Previous diagnosis of mental retardation
* Nitroglycerin use
* Asthma diagnosis, verified and treated by a primary care doctor
* Use of any other medication that may interact with the study medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: NAC 1st Trial, Placebo 2nd Trial: Group A first receives the commercially available sustained release form of NAC, then the matching placebo capsules both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days).
- Group B: Placebo 1st Trial, NAC 2nd Trial: Group B first receives the matching placebo capsules both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days , then receives commercially available sustained release form of NAC for the same period (8 total doses over 5 days).
Period: Randomization
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Initial Assessment
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: First Crossover
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Started | 12 | 11
Completed | 11 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Crossover
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Started | 11 | 11
Completed | 10 | 9
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Participants: This is the overall group of trial participants prior to randomization to either of the two crossover arms in the study.
Arm/Group | Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.64 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: BACS Composite RAW Score
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is an instrument that assesses the aspects of cognition found to be most impaired and most strongly correlated with outcome in patients with schizophrenia.
  The BACS composite raw score the total of the raw scores for the 6 subtests of the BACS (Verbal memory, token motor, digit sequencing, verbal fluency, symbol coding and executive functioning). The range, so we could be from 0-435. A high score total score is more favorable and indicates a higher level of cognition.
  The BACS requires less than 35 min to complete in patients with schizophrenia, yields a high completion rate in these patients, and has high reliability. The BACS was found to be as sensitive to cognitive impairment in patients with schizophrenia as a standard battery of tests that required over 2 h to administer. It is the raw sum of the test items and higher scores are favorable.
Time Frame: Baseline
Population: Subjects analyzed are those with complete data at baseline prior to dropout from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: This is the combined intervention group (both those receiving the intervention first and those receiving the intervention second).
- Placebo: This is the combined placebo group (both those receiving the placebo first and those receiving the placebo second).
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 229.04 (38.95) | 227.83 (44.44)

2. Primary Outcome: BACS Composite RAW Score
Description: as for outcome 1
Time Frame: Follow Up (5 days)
Population: Subjects analyzed are those with complete data at follow up and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale | 234.90 (35.15) | 237.77 (41.37)

3. Primary Outcome: BACS Composite RAW Score
Description: as for outcome 1
Time Frame: Change from Baseline at Follow Up (5 days)
Population: Subjects analyzed are only those with complete data at baseline and 5 day follow up in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale | -7.00 (13.89) | -5.59 (13.63)

4. Primary Outcome: BACS Composite RAW Score
Description: as for outcome 1
Time Frame: Baseline 1st Leg of Crossover
Population: Subjects analyzed are those with complete data at baseline prior to dropout from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group A: NAC 1st Trial, Placebo 2nd Trial: Group A first receives the commercially available sustained release form of NAC, then the matching placebo capsules both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days.
- Group B: Placebo 1st Trial, NAC 2nd Trial: Group B first receives the placebo and the receives rge commercially available sustained release form of NAC, in each arm the capsules both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days.
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 222.75 (40.72) | 226.45 (34.73)

5. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: Letter Number Sequencing (LNS) is a brief, standardized executive function task used to assess verbal working memory performance. The test involves a 24-item Experimental Condition, in which participants are read a series of letters and numbers and asked to recite both back in ascending order, with the numbers first and then the letters. Participants receive one point for each correct answer for a range of 0-24. Higher scores are better.
Time Frame: Baseline
Population: All participants were analyzed that had baseline data collected (including any that did not complete the time frame).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: This is the combined placebo/control group (both those receiving the placebo first and those receiving the placebo second).
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 13.43 (2.76) | 13.22 (3.15)

6. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: as for outcome 5
Time Frame: Follow Up (5 days)
Population: Subjects analyzed are those with complete data at follow up and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale | 13.48 (3.15) | 13.81 (3.49)

7. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: as for outcome 5
Time Frame: Change from Baseline at Follow Up (5 days)
Population: Subjects analyzed are those with complete data at follow up and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale | 0.14 (1.82) | -0.45 (2.36)

8. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: as for outcome 5
Time Frame: Baseline 1st Leg of Crossover
Population: Subjects analyzed are those with complete data at baseline prior to dropout from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group B: Placebo 1st Trial, NAC 2nd Trial: Group B first receives the placebo and then receives the commercially available sustained release form of NAC. Both are administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days).
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 13.33 (2.84) | 13.00 (3.35)

9. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: as for outcome 5
Time Frame: Follow Up 1st Leg of Crossover (5 Days)
Population: Subjects analyzed are those with complete data at follow up and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 12.75 (2.41) | 13.36 (3.67)

10. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: as for outcome 5
Time Frame: Baseline 2nd Leg of Crossover
Population: Subjects analyzed are those with complete data at 2nd baseline in the crossover and could include those that had dropped from the study if data was collected prior to drop out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 13.42 (3.08) | 13.55 (2.81)

11. Secondary Outcome: Letter/Number Sequencing Task Tests for Attention, Concentration & Mental Control (LNS) RAW SCORE.
Description: as for outcome 5
Time Frame: Follow Up 2nd Leg of Crossover (5 Days)
Population: Subjects analyzed are those with complete data at 2nd follow up in the crossover and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 11 | 9
units on a scale | 14.27 (3.41) | 14.44 (1.51)

12. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: Brief Visuospatial Memory Test (BVMT) is a measure of visuospatial memory. This task includes three trials of six geometric figures printed in a 2 x 3 array on separate pages. The respondent views the stimulus page for 10 seconds and is asked to draw as many of the figures as possible in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Scoring is based on accuracy of the figure as well as its location on the page. A range of 0-12 per trial is possible(0-36 total). Higher scores are better.
Time Frame: Baseline
Population: All participants were analyzed that had baseline data collected (including any that did not complete the time frame).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 20.35 (6.29) | 20.65 (7.87)

13. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: as for outcome 12
Time Frame: Follow Up (5 days)
Population: Subjects analyzed are those with complete data at follow up in the crossover and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Group A first receives the commercially available sustained release form of NAC, then the matching placebo capsules both administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days.
- Placebo: Group B first receives the placebo and then receives the commercially available sustained release form of NAC. Both are administered at 1200mg twice a day for 3 full days, along with 1200mg once on the evening prior to and once on the morning following the 3 days (8 total doses over 5 days).
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale | 17.90 (6.29) | 17.68 (5.86)

14. Primary Outcome: BACS Composite RAW Score
Description: as for outcome 1
Time Frame: Follow Up 1st Leg of Crossover (5 Days)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 231.58 (43.25) | 237.00 (37.62)

15. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: as for outcome 12
Time Frame: Change from Baseline at Follow Up (Baseline - Follow Up)
Population: Subjects analyzed are those with complete data at all timepoints and does not include those that had dropped from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale | 2.57 (5.13) | 2.77 (5.76)

16. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: as for outcome 12
Time Frame: Baseline 1st Leg of Crossover
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 20.67 (5.82) | 19.73 (16.55)

17. Primary Outcome: BACS Composite RAW Score
Description: as for outcome 1
Time Frame: Baseline 2nd Leg of Crossover
Population: Subjects analyzed are those with complete data at baseline prior to dropout from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 229.08 (53.38) | 235.91 (239.33)

18. Primary Outcome: BACS Composite RAW Score
Description: as for outcome 1
Time Frame: Follow Up 2nd Leg of Crossover (5 Days)
Population: Subjects analyzed are those with complete data at follow up and does not include those dropped out from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 11 | 9
units on a scale | 238.55 (46.67) | 239.33 (21.85)

19. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: as for outcome 12
Time Frame: Follow Up 1st Leg of Crossover (5 Days)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 16.55 (6.07) | 18.25 (7.39)

20. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: as for outcome 12
Time Frame: Baseline 2nd Leg of Crossover
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 11
units on a scale | 21.50 (7.80) | 20.00 (7.01)

21. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) RAW SCORE.
Description: as for outcome 12
Time Frame: Follow Up 2nd Leg of Crossover (5 Days)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 11 | 9
units on a scale | 18.82 (5.69) | 17.44 (4.85)

22. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)Total Score
Description: Brief Psychiatric Rating Scale (BPRS) utilized before and after treatment. BPRS total score is a total of the 18 item scores with a range of 18-126. It is used to measure schizophrenia symptoms and to assess change in them over time. There are 18 symptom sub scores. Each symptom is rated 1-7 (not present to extremely severe) and then all items are summed for the total score. Higher scores indicate more severe symptoms.
  The BPRS is the gold-standard overall measure of schizophrenia symptoms which will be utilized to demonstrate that the intervention does not cause worsening of the illness symptoms apart from the usual fluctuations of the natural course.
Time Frame: Pre Screening
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 12 | 12
units on a scale | 30.92 (7.20) | 28.41 (7.41)

23. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)Total Score
Description: as for outcome 22
Time Frame: End of Trial
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 10 | 9
units on a scale | 32.80 (7.31) | 27.78 (8.91)

24. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)Total Score
Description: as for outcome 22
Time Frame: Change from PreScreening at End of Trial
Population: Analyses only used matched cases and does not include participants with incomplete data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: NAC 1st Trial, Placebo 2nd Trial | Group B: Placebo 1st Trial, NAC 2nd Trial
Number analyzed (Participants) | 10 | 9
units on a scale | 1.70 (2.36) | 0.89 (1.05)

ADVERSE EVENTS:
Groups:
- Placebo: First Crossover Follow Up: This group of participants received the placebo on the first day in the crossover design.
- NAC: First Crossover Follow Up: This group of participants received the active treatment (NAC) on the first day of the crossover study.
- Placebo: Second Crossover Follow Up: This group of participants received the placebo on the second day in the crossover design.
- NAC: Second Crossover Follow Up: This group of participants received the active treatment (NAC) on the second day of the crossover study.
Arm/Group | Placebo: First Crossover Follow Up | NAC: First Crossover Follow Up | Placebo: Second Crossover Follow Up | NAC: Second Crossover Follow Up
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/11 | 6/12 | 4/11 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: First Crossover Follow Up (N=11) | NAC: First Crossover Follow Up (N=12) | Placebo: Second Crossover Follow Up (N=11) | NAC: Second Crossover Follow Up (N=11)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Appetite Loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight Gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Libido Increase (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep Disturbance (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Memory Loss (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal Congestion (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizzyness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes